CLINICAL TRIAL: NCT04133545
Title: Discontinuation for Oral Anticoagulants During the First Year of Use in Patients With Atrial Fibrillation Covered by a Medical Insurance
Brief Title: Discontinuation for Oral Anticoagulants in Patients With Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, JOSE LUIS CARLOS NAVARRO, MD, Hospital Italiano de Buenos Aires
Other Study IDs: Protocol_3525
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Auricular Fibrillation; Anticoagulant Drugs
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DOAC: Direct oral anticoagulant
- OAC: Vitamin K anticoagulant

SUMMARY:
The purpose of this study is to compare the discontinuation rates for vitamin K antagonists and for direct oral anticoagulants during their first year

DETAILED DESCRIPTION:
The purpose of this study is to compare the discontinuation rates for vitamin K antagonists and for direct oral anticoagulants during their first year of use after their initiation during hospitalization in patients covered by our health insurance plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years of age covered by our Health Care Insurance Plan.
2. Indication for oral anticoagulation with an expected duration of use of no less than 1 year.

Exclusion Criteria:

1. Refusal to take part.
2. Use of oral anticoagulants within 6 months prior to admission.
3. Presence of mechanical prosthetic valve.
4. Chronic renal failure with creatinine clearance <30 mL/min (estimated using the MDRD formula).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients belonging to a Health Management Organization suffering from atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Anticoagulant Discontinuation Rate | One year
  Anticoagulant Discontinuation Rate

SECONDARY OUTCOMES:
Discontinuation Predictors | One year
  Discontinuation Predictors

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Navarrro Estrada, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No